CLINICAL TRIAL: NCT05368363
Title: Accuracy of Preoperative Evaluation of Inferior Vena Cava Collapsibility Index and Caval Aorta Index for Prediction of Hypotension After Induction of General Anaesthesia: "A Prospective Observational Study"
Brief Title: Inferior Vena Cava Collapsibility Index and Caval Aorta Index for Prediction of Hypotension General Anaesthesia
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Omar Ahmed, Associate professor of Anesthesia, pain management & surgical ICU, Cairo University
Other Study IDs: MD-266-2020
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: IVC Collapsibility Index as Predictor for Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To estimate sensitivity and specificity of preoperative IVCCI, max aortic diameter and IVC:Ao index as predictors of hypotension after induction of general anesthesia.
2. To compare accuracy of preoperative values of IVC: Ao index to preoperative IVCCI in prediction of hypotension after induction of general anesthesia.

DETAILED DESCRIPTION:
After obtaining approval from the hospital ethics committee, informed consent will be obtained from 102 patients who will undergo elective surgery requiring general anaesthesia in supine position. Patients will be evaluated by history taking and proper examination. Pre-operative investigations will be checked. On the day of surgery, pre-operative fasting for 8 hours will be confirmed.

Upon arrival to the operating room, routine monitors in the form of pulse oximetry, electrocardiogarm and non-invasive blood pressure monitors will be applied. Intravenous line will be secured and routine premedications (ranitidine 50 mg and ondansetron 4 mg) will be administered.

1. IVC Ultrasonography (IVCCI and IVC:Ao index) :

   While the patient is lying supine, the IVC and aorta will be examined before induction of general anaesthesia using a curved ultrasound transducer set to abdominal mode with a B-mode scan (1-5 MHz; Acuson x300; Siemens Healthcare, Seoul, Korea).

   The transducer is placed in the subxiphoid region in a longitudinal position. IVC measurements are made just distal to the IVC-hepatic vein junction, approximately 3 to 4 cm distal to the right atrium. The IVC is identified by Doppler waveform, compressibility and phasic collapse with respiration. The maximum (IVCDmax) and minimum (IVCDmin) internal anteroposterior (AP) diameters of the IVC at the end of expiration and inspiration respectively over the same respiratory cycle will be measured. The IVCCI is derived from the equation: (7) IVCCI = [ (IVCDmax - IVCDmin) / IVCDmax ] X 100. To the left of the IVC, the abdominal aorta is visualized 10 mm above the coeliac trunk. The maximum internal AP diameter of the abdominal aorta is measured during systole. The IVC:Ao index is derived by taking the ratio of the maximum IVC diameter during expiration and the maximal abdominal aortic diameter during systole.
2. Induction of anesthesia:

Standard noninvasive monitoring including ECG, noninvasive blood pressure (BP) measurements every minute and oxygen saturation will be applied. Heart rate (HR), SBP and MBP will be recorded immediately before general anaesthesia and will be defined as baseline readings.

General anaesthesia induction will be started using propofol intravenous anaesthetic (2 mg/kg) and Fentanyl (1 microgram/kg) and Atracrurium non-depolarizing muscle relaxant (0.5 mg/kg).Smooth endotracheal intubation with appropriate sized-cuffed endotracheal tube will be done after 3 mins of manual bag mask ventilation. Confirmation of endotracheal intubation will be done by 3 successive capnography waves and by bilateral lung auscultation. Meanwhile, the noninvasive BP will be recorded immediately after induction, then 5 and 10 minutes post induction, with continuous monitoring of other vital parameters (HR and oxygen saturation) during the postinduction period.

Any episode of hypotension (defined as mean arterial pressure < 80% of the baseline reading or or MAP less than 60 mmHg) will be managed by ephedrine 5 mg every 2 min to increase SBP to 80% of the baseline or MAP more than 70 mmHg. If the hypotensive episode persisted for 2 minutes, another bolus of norepinephrine will be administered. Any episodes of bradycardia (defined as heart rate less than 50 bpm) will be managed by atropine (0.01 mg/kg).

Patients will then be divided into two groups depending on whether they'll develop post general anesthesia induction hypotension or won't. Any complications, such as hypoxia or allergic reaction will be noted and managed accordingly.

The attending anesthesiologist who will perform the induction of general anaesthesia and monitor the patient during the study period will be blinded to the ultrasound measurements of IVCCI and IVC :Ao index recorded pre-operatively.

Measurement tools

* Mean arterial blood pressure will be measured in supine position in one of the upper limbs in the operating room at 1-minute intervals starting from the baseline preoperative reading until skin incision as follows: 1-minute post-induction reading, 2-minutes post-induction reading, pre-intubation reading & post-intubation readings until skin incision. Taking in consideration that the maximum time for recording the readings of the blood pressure is 15 minutes because if hypotension occurred after this time it is unlikely to be due to the effect of induction of anesthesia.
* Heart rate will be recorded at 1-minute intervals starting from the baseline pre-operative reading until skin incision as follows: 1-minute post-induction reading, 2-minutes post-induction reading, pre-intubation reading & post-intubation readings until skin incision.
* Demographic data: (age - gender - comorbidities - current medications).
* The incidence of post-induction hypotension.
* The incidence of bradycardia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 60 years old
* Patients undergoing elective surgery under general anesthesia.
* ASA I, II

Exclusion Criteria:

* Patients with BMI more than 35.
* Pregnant patients
* Emergency cases
* Patients with a baseline arterial SBP less than 90 mmHg or mean arterial pressure (MAP) less than 70 mmHg.
* Patients with major severe vascular disease, Unstable angina, Ejection fraction< 40 %, Respiratory distress, Implanted pacemaker or Patients on angiotensin converting enzyme inhibitors or angiotensin receptor blockers
* Patients with increased intra-abdominal pressure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18 - 60 years old , Patients undergoing elective surgery under general anesthesia, ASA I, II
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Area under receiver operating characteristic curves (AUROC) of the preoperative IVCCI inprediction of post-induction hypotension | 5 minutes
  Area under receiver operating characteristic curves (AUROC) of the preoperative IVCCI inprediction of post-induction hypotension

SECONDARY OUTCOMES:
Correlation between each of maximum aortic diameter with the percentage of themaximum decrease in mean arterial pressure after induction of anesthesia | 5 minutes
  Correlation between each of maximum aortic diameter with the percentage of themaximum decrease in mean arterial pressure after induction of anesthesia
Correlation between each of IVC collapsibility index with the percentage of themaximum decrease in mean arterial pressure after induction of anesthesia | 5 minutes
  Correlation between each of IVC collapsibility index with the percentage of themaximum decrease in mean arterial pressure after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Heba Omar, Study Director — associate professor of anesthesia and surgical ICU, faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910
- [Background] Salama ER, Elkashlan M. Pre-operative ultrasonographic evaluation of inferior vena cava collapsibility index and caval aorta index as new predictors for hypotension after induction of spinal anaesthesia: A prospective observational study. Eur J Anaesthesiol. 2019 Apr;36(4):297-302. doi: 10.1097/EJA.0000000000000956. PMID 30664523